CLINICAL TRIAL: NCT00631293
Title: Study on the Effect of Lactisole on the Intestinal Glucose Uptake
Brief Title: Study of the Effect of Lactisole on the Intestinal Glucose Uptake
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: VIB (Unknown)
Responsible Party: Dirk Iserentant, PhD, University Ghent
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2008/103
Record Dates: First submitted 2008-02-26; First posted 2008-03-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — lactisole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): administration of lactisole
  Interventions: Dietary Supplement: lactisole
- 2 (Placebo Comparator): administration of placebo
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: lactisole — administration of lactisole followed by placebo
  Arms: 1
Other: placebo — administration of placebo followed by lactisole
  Arms: 2

SUMMARY:
Study of the effect of lactisole on glucose uptake

ELIGIBILITY:
Inclusion Criteria:

* Male subject, between 18 and 50 years
* General good health condition

Exclusion Criteria:

* Overweight (Body Mass Index ≥30)
* Metabolic disorders
* History of gastrointestinal disorders
* Regular (daily) intake of medication
* Smoking more than 10 cigarettes/day
* History of drug abuse
* Exhaustive (> 3 units/day) alcohol consumption
* Exhaustive (> 5 units/day) caffeine consumption (coffee, tea, cola, or other caffeine based drinks)
* Recent (in the last 14 days) donation of blood
* Recent (in the last 2 days) donation of blood plasma
* Participation in another trial within 4 weeks before the start of the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Differences in glucose uptake rate in lactisole treated subjects versus placebo treated subjects during oral glucose tolerance test | 5 weeks

SECONDARY OUTCOMES:
Differences in blood insulin, glucagon, triglycerides, GIP and GLP-1 in lactisole treated subjects versus placebo treated subjects during oral glucose tolerance test, ECG | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luc Van Bortel, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium